CLINICAL TRIAL: NCT01302041
Title: A Phase 2, Open-label, Single-arm, Efficacy and Safety Study of Enzalutamide (MDV3100) in Patients With Hormone-naïve Prostate Cancer
Brief Title: A Study to Test if Enzalutamide is Effective and Safe in Prostate Cancer Patients Who Have Never Had Hormone Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9785-CL-0321; 2010-021287-16 (EudraCT Number)
Record Dates: First submitted 2011-02-21; First posted 2011-02-23 (Estimated); Results first posted 2016-04-06 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-05

CONDITIONS: Prostate Cancer
Keywords: bone turnover; hormone-naïve; prostate specific antigen; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Enzalutamide (Experimental): Participants received oral enzalutamide at 160 mg once daily for 24 weeks. Participants who had clinical benefit at Week 25 could continue to receive enzalutamide until disease progression, objective or clinical, or occurrence of an unacceptable toxicity, at the discretion of the investigator.
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Enzalutamide — Oral
  Other Names: Xtandi; MDV3100

SUMMARY:
To evaluate the effect of enzalutamide on prostate specific antigen (PSA) level in men with prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate cancer (all stages) for whom androgen deprivation therapy is indicated (except when indicated in a neoadjuvant/adjuvant therapy)
* Asymptomatic from prostate cancer
* Non-castrate level of testosterone (≥ 8 nmol/L (230 ng/dL)) at screening
* PSA ≥ 2 ng/mL at screening

Exclusion Criteria:

Has previously or is currently receiving:

* Hormonal therapy with intent to treat prostate cancer
* Systemic glucocorticoids
* Chemotherapy with the intent to treat prostate cancer
* Opiate analgesics for pain from prostate cancer
* Radiation therapy for treatment of the primary tumor or metastases
* Has history of known or suspected brain or skull metastases or leptomeningeal disease
* Has history of seizure including febrile seizure or any condition that may predispose to seizure or history of loss of consciousness or transient ischemic attack
* Clinically significant cardiovascular disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2011-05-06 (Actual); Primary Completion 2012-07-29 (Actual); Study Completion 2017-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Europe B.V.
Locations (12):
- Belgium (4):
  - Site BE1003, Brussels
  - Site BE1001, Brussels
  - Site BE1002, Kortrijk
  - Site BE1005, Leuven
- Czechia (2):
  - Site CZ3006, Olomouc
  - Site CZ3002, Prague
- Denmark (3):
  - Site DK4001, Aarhus N
  - Site DK4004, Copenhagen
  - Site DK4002, Herlev
- Germany (3):
  - Site DE5005, Aachen
  - Site DE5007, Bonn
  - Site DE5003, Hanover

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Trump D. Commentary on: "Enzalutamide monotherapy in hormone-naive prostate cancer: primary analysis of an open-label, single-arm, phase 2 study." Tombal B, Borre M, Rathenborg P, Werbrouck P, Van Poppel H, Heidenreich A, Iversen P, Braeckman J, Heracek J, Baskin-Bey E, Ouatas T, Perabo F, Phung D, Hirmand M, Smith MR. Institut de Recherche Clinique, Universite Catholique de Louvain, Brussels, Belgium. Electronic address: bertrand.tombal@uclouvain.be. Aarhus University Hospital, Aarhus, Denmark. Herlev Hospital, Herlev, Denmark. AZ Groeninge Kortrijk, Kortrijk, Belgium. UZ Leuven, Leuven, Belgium. Klinik und Poliklinik fur Urologie, RWTH University Aachen, Aachen, Germany. Rigshospitalet, University of Copenhagen, Copenhagen, Denmark. UZ Brussel, Brussels, Belgium. Univerzita Karlova v Praze, Prague, Czech Republic. Astellas Pharma Global Development, Leiden, Netherlands. Astellas Pharma Global Development, Northbrook, IL, USA. Medivation Inc, San Francisco, CA, USA. Massachusetts General Hospital Cancer Center, Boston, MA, USA: Lancet Oncol. 2014 May;15(6):592-600; doi: 10.1016/S1470-2045(14)70129-9. [Epub 2014 Apr 14]. Urol Oncol. 2016 May;34(5):248-9. doi: 10.1016/j.urolonc.2015.03.012. Epub 2015 Apr 30. PMID 25937426
- [Derived] Tombal B, Borre M, Rathenborg P, Werbrouck P, Van Poppel H, Heidenreich A, Iversen P, Braeckman J, Heracek J, Baskin-Bey E, Ouatas T, Perabo F, Phung D, Baron B, Hirmand M, Smith MR. Long-term Efficacy and Safety of Enzalutamide Monotherapy in Hormone-naive Prostate Cancer: 1- and 2-Year Open-label Follow-up Results. Eur Urol. 2015 Nov;68(5):787-94. doi: 10.1016/j.eururo.2015.01.027. Epub 2015 Feb 14. PMID 25687533
- [Derived] Tombal B, Borre M, Rathenborg P, Werbrouck P, Van Poppel H, Heidenreich A, Iversen P, Braeckman J, Heracek J, Baskin-Bey E, Ouatas T, Perabo F, Phung D, Hirmand M, Smith MR. Enzalutamide monotherapy in hormone-naive prostate cancer: primary analysis of an open-label, single-arm, phase 2 study. Lancet Oncol. 2014 May;15(6):592-600. doi: 10.1016/S1470-2045(14)70129-9. Epub 2014 Apr 14. PMID 24739897
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=44

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multinational, phase 2, open-label, single-arm, efficacy and safety study of oral enzalutamide in participants with prostate cancer who had noncastrate levels of testosterone at study entry.
Pre-assignment Details: Eighty-two participants were assessed for participation in the study, 15 were excluded and 67 were enrolled. Participants who continued to receive clinical benefit as assessed by the investigator and did not meet any treatment discontinuation criteria were eligible to transition to an open-label extension study 9785-CL-0123 (NCT02960022).
Period: Overall Study
Arm/Group | Enzalutamide
Started | 67
Treatment Received | 67
Completed | 27 (Participants who discontinued treatment and completed the 30-day follow-up visit)
Not Completed | 40
Not completed — Death | 5
Not completed — Withdrawal by Subject | 4
Not completed — Other-Transitioned to 9785-CL-0123 | 29
Not completed — Other-Miscellaneous Reason | 2

BASELINE CHARACTERISTICS:
Arm/Group | Enzalutamide
Number analyzed (Participants) | 67
Age, Continuous [Median (Full Range); unit: Years] | 73.0 [48 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 67
Body Mass Index (BMI) [Median (Full Range); unit: kg/m²] | 26.17 [20.8 to 39.7]
Prostate Specific Antigen (PSA) [Median (Inter-Quartile Range); unit: ng/mL] | 18.2 (102.990) [6.4 to 45.0]
Duration of Prostate Cancer [Median (Full Range); unit: years] | 1.0 [0 to 16]
Total Gleason Score at Initial Diagnosis [Count of Participants; unit: Participants] — A system of grading prostate cancer tissue based on how it looks under a microscope. Gleason scores range from 2 to 10 and indicate how likely it is that a tumor will spread. A low Gleason score means the cancer tissue is similar to normal prostate tissue and the tumor is less likely to spread; a high Gleason score means the cancer tissue is very different from normal and the tumor is more likely to spread.
  Participants
    4 | 1
    5 | 5
    6 | 10
    7 | 34
    8 | 7
    9 | 6
    10 | 3
    Unknown | 1
Clinical Tumor Stage (T) at Initial Diagnosis [Count of Participants; unit: Participants]
  TX: Primary tumor cannot be assessed | 1
  T0: No evidence of primary tumor | 1
  T1: Tumor neither palpable or visible by imaging | 9
  T2: Tumor confined within the prostate | 31
  T3: Tumor extends through the prostatic capsule | 18
  T4: Tumor is fixed or invades adjacent structures | 1
  Unknown | 6
Clinical Lymph Node Stage (N) at Initial Diagnosis [Count of Participants; unit: Participants]
  NX: Regional lymph nodes were not assessed | 24
  N0: No regional lymph node metastasis | 22
  N1: Metastasis in regional lymph node(s) | 6
  Unknown | 15
Distant Metastasis (M) at Initial Diagnosis [Count of Participants; unit: Participants]
  MX: Distant metastasis could not be assessed | 11
  M0: No distant metastasis | 35
  M1: Distant metastasis | 10
  Unknown | 11
Participants With Metastases at Study Entry [Count of Participants; unit: Participants] | 26
Number of Metastatic Lesions by Bone Scan [Median (Full Range); unit: Lesions] | 1 [1 to 8]
Previous Interventions [Count of Participants; unit: Participants] — Participants may have received more than one intervention
  Participants
    Radiotherapy | 16
    Prostatectomy | 24
    Transurethral Resection of the Prostate | 4
    Pelvic Lymph Node Dissection | 6
    Watchful Waiting | 14
    Other Surgeries/Procedures | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Prostate-Specific Antigen (PSA) Response at Week 25
Description: A PSA response was defined as a decline from Baseline in PSA level of 80% or greater. Blood samples for PSA were collected and analyzed at a central laboratory. Participants with an unknown or missing response or who discontinued prior to week 25 for any reason were treated as non-responders.
Time Frame: Baseline and Week 25
Population: The analysis population was safety analysis set (SAF), which consisted of participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Enzalutamide
Number analyzed (Participants) | 67
Percentage of Participants | 92.5 [83.44 to 97.53]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Each adverse event (AE) was assessed by the investigator for causal relationship to the study drug; those deemed possibly or probably related to study drug are reported as drug regimen related AEs (DRRAEs).
  A serious adverse event (SAE) was defined as any untoward medical occurrence that at any dose:
  * Resulted in death
  * Was life-threatening
  * Resulted in persistent or significant disability/incapacity
  * Resulted in congenital anomaly or birth defect
  * Required inpatient hospitalization or led to prolongation of hospitalization
  * Other medically important events.
Time Frame: From first dose of study drug up to 30 days after last dose of study drug; median duration of treatment of 1666.0 days (range of 52-2052)
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide
Number analyzed (Participants) | 67
Participants
  Any Adverse Events | 67
  Drug Regimen Related Adverse Events | 65
  Deaths | 5
  Serious Adverse Events | 24
  Drug Regimen Related Serious Adverse Events | 5
  AEs Leading to Discontinuation of Study Drug | 14
  DRRAEs Leading to Discontinuation of Study Drug | 7

3. Secondary Outcome: Percent Change From Baseline in PSA
Time Frame: Baseline and Weeks 25, 49, 97, 169 and Week 265 (End of Study)
Population: Safety Analysis Set with available data at each time point
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Enzalutamide
Number analyzed (Participants) | 67
Percent Change
  Week 25: number analyzed (Participants) | 63
  Week 25 | -97.82 (5.744)
  Week 49: number analyzed (Participants) | 54
  Week 49 | -98.96 (2.767)
  Week 97: number analyzed (Participants) | 45
  Week 97 | -99.44 (1.114)
  Week 169: number analyzed (Participants) | 42
  Week 169 | -91.74 (27.808)
  Week 265 (End of Study): number analyzed (Participants) | 27
  Week 265 (End of Study) | -0.70 (368.253)

4. Secondary Outcome: Percent Change From Baseline in Sex Hormone-Binding Globulin (SHBG)
Time Frame: Baseline and Weeks 25 and 49
Population: Safety Analysis Set with available data at each time point
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Enzalutamide
Number analyzed (Participants) | 67
Percent Change
  Week 25: number analyzed (Participants) | 59
  Week 25 | 100.60 (49.362)
  Week 49: number analyzed (Participants) | 53
  Week 49 | 88.45 (41.911)

5. Secondary Outcome: Percent Change From Baseline in Androstenedione
Time Frame: Baseline and Weeks 25 and 49
Population: Safety Analysis Set with available data at each time point
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Enzalutamide
Number analyzed (Participants) | 67
Percent Change
  Week 25: number analyzed (Participants) | 61
  Week 25 | 51.06 (59.367)
  Week 49: number analyzed (Participants) | 51
  Week 49 | 49.94 (55.449)

6. Secondary Outcome: Percent Change From Baseline in Dehydroepiandrosterone (DHEA)
Time Frame: Baseline and Weeks 25 and 49
Population: Safety Analysis Set with available data at each time point
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Enzalutamide
Number analyzed (Participants) | 67
Percent Change
  Week 25: number analyzed (Participants) | 62
  Week 25 | 9.59 (58.247)
  Week 49: number analyzed (Participants) | 51
  Week 49 | 10.54 (54.864)

7. Secondary Outcome: Percent Change From Baseline in Dihydrotestosterone (DHT)
Time Frame: Baseline and Week 25 and 49
Population: Safety Analysis Set with available data at each time point
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Enzalutamide
Number analyzed (Participants) | 67
Percent Change
  Week 25: number analyzed (Participants) | 61
  Week 25 | 51.72 (57.511)
  Week 49: number analyzed (Participants) | 45
  Week 49 | 74.35 (101.451)

8. Secondary Outcome: Percent Change From Baseline in Estradiol
Time Frame: Baseline and Weeks 25 and 49
Population: Safety Analysis Set with available data at each time point
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Enzalutamide
Number analyzed (Participants) | 67
Percent Change
  Week 25: number analyzed (Participants) | 59
  Week 25 | 71.69 (73.150)
  Week 49: number analyzed (Participants) | 52
  Week 49 | 81.00 (82.811)

9. Secondary Outcome: Percent Change From Baseline in Follicle-Stimulating Hormone (FSH)
Time Frame: Baseline and Weeks 25 and 49
Population: Safety Analysis Set with available data at each time point
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Enzalutamide
Number analyzed (Participants) | 67
Percent Change
  Week 25: number analyzed (Participants) | 58
  Week 25 | 46.99 (46.389)
  Week 49: number analyzed (Participants) | 52
  Week 49 | 62.18 (78.371)

10. Secondary Outcome: Percent Change From Baseline in Luteinizing Hormone (LH)
Time Frame: Baseline and Weeks 25 and 49
Population: Safety Analysis Set with available data at each time point
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Enzalutamide
Number analyzed (Participants) | 67
Percent Change
  Week 25: number analyzed (Participants) | 58
  Week 25 | 184.66 (120.683)
  Week 49: number analyzed (Participants) | 52
  Week 49 | 215.18 (163.732)

11. Secondary Outcome: Percent Change From Baseline in Prolactin
Time Frame: Baseline and Weeks 25 and 49
Population: Safety Analysis Set with available data at each time point
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Enzalutamide
Number analyzed (Participants) | 67
Percent Change
  Week 25: number analyzed (Participants) | 60
  Week 25 | 16.79 (45.497)
  Week 49: number analyzed (Participants) | 53
  Week 49 | 9.64 (30.003)

12. Secondary Outcome: Percent Change From Baseline in Total Testosterone
Time Frame: Baseline and Weeks 25 and 49
Population: Safety Analysis Set with available data at each time point
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Enzalutamide
Number analyzed (Participants) | 67
Percent Change
  Week 25: number analyzed (Participants) | 63
  Week 25 | 114.29 (73.692)
  Week 49: number analyzed (Participants) | 51
  Week 49 | 101.73 (76.070)

13. Secondary Outcome: Percent Change From Baseline in Free Testosterone
Time Frame: Baseline and Weeks 25 and 49
Population: Safety Analysis Set with available data at each time point
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Enzalutamide
Number analyzed (Participants) | 67
Percent Change
  Week 25: number analyzed (Participants) | 60
  Week 25 | 46.39 (59.551)
  Week 49: number analyzed (Participants) | 51
  Week 49 | 43.74 (55.721)

14. Secondary Outcome: Plasma Concentration of Enzalutamide at Pre-dose (Ctrough)
Time Frame: Pre-dose at Weeks 2, 3, 4, 5, 9, 13, 21 and 25
Population: Pharmacokinetic Analysis Set (PKAS) (participants who had taken at least 1 dose of study drug and who had at least 1 pharmacokinetic concentration value) with available data at each time point
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Enzalutamide
Number analyzed (Participants) | 67
μg/mL
  Week 2: number analyzed (Participants) | 61
  Week 2 | 7.225 (1.8050)
  Week 3: number analyzed (Participants) | 66
  Week 3 | 10.559 (2.1967)
  Week 4: number analyzed (Participants) | 62
  Week 4 | 11.838 (2.4605)
  Week 5: number analyzed (Participants) | 65
  Week 5 | 12.161 (2.8496)
  Week 9: number analyzed (Participants) | 63
  Week 9 | 11.606 (3.0084)
  Week 13: number analyzed (Participants) | 63
  Week 13 | 11.868 (2.9760)
  Week 21: number analyzed (Participants) | 62
  Week 21 | 11.224 (2.8899)
  Week 25: number analyzed (Participants) | 63
  Week 25 | 11.668 (2.7624)

15. Secondary Outcome: Plasma Concentration of Enzalutamide Metabolite M2 at Pre-dose (Ctrough)
Time Frame: Pre-dose at Weeks 2, 3, 4, 5, 9, 13, 21 and 25
Population: Pharmacokinetic Analysis Set with available data at each time point
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Enzalutamide
Number analyzed (Participants) | 67
μg/mL
  Week 2: number analyzed (Participants) | 61
  Week 2 | 2.527 (1.0440)
  Week 3: number analyzed (Participants) | 66
  Week 3 | 5.344 (1.7079)
  Week 4: number analyzed (Participants) | 62
  Week 4 | 8.182 (2.4366)
  Week 5: number analyzed (Participants) | 65
  Week 5 | 9.962 (2.7584)
  Week 9: number analyzed (Participants) | 63
  Week 9 | 12.128 (3.1262)
  Week 13: number analyzed (Participants) | 63
  Week 13 | 12.780 (3.2564)
  Week 21: number analyzed (Participants) | 62
  Week 21 | 11.717 (2.9502)
  Week 25: number analyzed (Participants) | 63
  Week 25 | 12.146 (2.5845)

16. Secondary Outcome: Percentage of Participants With a PSA Response at Weeks 49, 97 and 169
Description: A PSA response was defined as a decline from baseline in PSA level of 80% or greater. Blood samples for PSA were collected and analyzed at a central laboratory. Participants with an unknown or missing response or who discontinued prior to week 49, week 97 or week 169 for any reason were treated as non-responders.
Time Frame: Baseline and Weeks 49, 97 and 169
Population: Safety Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Enzalutamide
Number analyzed (Participants) | 67
Percentage of Participants
  Week 49 | 80.6 [69.11 to 89.24]
  Week 97 | 67.2 [54.60 to 78.15]
  Week 169 | 56.7 [44.04 to 68.78]

17. Secondary Outcome: Percentage of Participants With a 90% or Greater Reduction From Baseline in PSA Level
Description: Participants with unknown or missing PSA results at week 25 or who discontinued prior to week 25 were considered non-responders at week 25. Participants with unknown or missing PSA results at week 49, week 97 or week 169 were considered non-responders.
Time Frame: Baseline and Weeks 25, 49, 97 and 169
Population: Safety Analysis Set; Week 49, 97 and 169 analyses include participants who were on study at each time point
Measure: Number; unit: Percentage of Participants
Arm/Group | Enzalutamide
Number analyzed (Participants) | 67
Percentage of Participants
  Week 25 | 91.0
  Week 49: number analyzed (Participants) | 54
  Week 49 | 98.1
  Week 97: number analyzed (Participants) | 45
  Week 97 | 100.0
  Week 169: number analyzed (Participants) | 42
  Week 169 | 88.1

18. Secondary Outcome: Percentage of Participants With PSA ≤ 4 ng/ml
Description: Participants with unknown or missing PSA results at week 25 or who discontinued prior to Week 25 were considered non-responders at Week 25. Participants with unknown or missing PSA results at week 49, 97 and 169 were considered non-responders.
Time Frame: Weeks 25, 49, 97 and 169
Population: Safety Analysis Set; Week 49, 97 and 169 analyses include participants who were on study at each time point
Measure: Number; unit: Percentage of Participants
Arm/Group | Enzalutamide
Number analyzed (Participants) | 67
Percentage of Participants
  Week 25 | 92.5
  Week 49: number analyzed (Participants) | 54
  Week 49 | 94.4
  Week 97: number analyzed (Participants) | 45
  Week 97 | 100.0
  Week 169: number analyzed (Participants) | 42
  Week 169 | 95.2

19. Secondary Outcome: Percentage of Participants With PSA ≤ 0.1 ng/ml
Description: Participants with unknown or missing PSA results at week 25 or who discontinued prior to week 25 were considered non-responders at week 25. Participants with unknown or missing PSA results at week 49, 97 or 169 were considered non-responders.
Time Frame: Weeks 25, 49, 97 and 169
Population: Safety Analysis Set; Week 49, 97 and 169 analyses include participants who were on study at each time point
Measure: Number; unit: Percentage of Participants
Arm/Group | Enzalutamide
Number analyzed (Participants) | 67
Percentage of Participants
  Week 25 | 44.8
  Week 49: number analyzed (Participants) | 54
  Week 49 | 63.0
  Week 97: number analyzed (Participants) | 45
  Week 97 | 73.3
  Week 169: number analyzed (Participants) | 42
  Week 169 | 61.9

20. Secondary Outcome: Maximum Decline From Baseline in PSA
Description: The maximum decline from Baseline in PSA was calculated as the largest reduction from Baseline in PSA level that occurred at any point after treatment start up to week 25 and up to and including the assessment made at the safety follow-up visit, divided by the PSA Baseline value and multiplied by 100, i.e., the maximum percent change from baseline.
Time Frame: Baseline to Week 25 and from Baseline up to the EOS date of 27 Apr 2017; median duration of treatment of 1666.0 days (range of 52-2052)
Population: Safety Analysis Set with available data at each time point
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Enzalutamide
Number analyzed (Participants) | 67
Percent Change
  Maximum Decline by Week 25 | -98.32 (2.880)
  Maximum Decline by EOS | -99.10 (2.659)

21. Secondary Outcome: Time to PSA Response
Description: Time to PSA response (PSA decline ≥ 80% from Baseline) is defined as the time interval from the first study drug dose to the first date a decline from Baseline in PSA level of 80% or greater was recorded. Time to response was estimated using the Kaplan-Meier method.
Time Frame: From first dose until the EOS date of 27-Apr-2017; median duration of treatment of 1666.0 days (range of 52-2052)
Population: Safety Analysis Set
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Enzalutamide
Number analyzed (Participants) | 67
Days | 29 [28 to 31]

22. Secondary Outcome: Time to PSA Decline ≥ 90%
Description: Time to PSA decline ≥ 90% is defined as the time interval from the first study drug dose to the first date a decline from Baseline in PSA level of 90% or greater was recorded. Time to PSA decline ≥ 90% was estimated using the Kaplan-Meier method.
Time Frame: From first dose until the EOS date of 27-Apr-2017; median duration of treatment of 1666.0 days (range of 52-2052)
Population: Safety Analysis Set
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Enzalutamide
Number analyzed (Participants) | 67
Days | 55 [29 to 57]

23. Secondary Outcome: Time to PSA ≤ 4 ng/ml
Description: Time to PSA ≤ 4 ng/ml is defined as the time interval from the first study drug dose to the first date a decline in PSA to a result of 4 ng/ml or below was recorded. Time to PSA ≤ 4 ng/ml was estimated using the Kaplan-Meier method.
Time Frame: From first dose until the EOS date of 27-Apr-2017; median duration of treatment of 1666.0 days (range of 52-2052)
Population: Safety Analysis Set
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Enzalutamide
Number analyzed (Participants) | 67
Days | 29 [9 to 57]

24. Secondary Outcome: Time to PSA ≤ 0.1 ng/ml
Description: Time to PSA ≤ 0.1 ng/ml is defined as the time interval from the first study drug dose to the first date a decline in PSA to a result of 0.1 ng/ml or below was recorded.
  Time to PSA ≤ 0.1 ng/ml was estimated using the Kaplan-Meier method.
Time Frame: From first dose until the EOS date of 27-Apr-2017; median duration of treatment of 1666.0 days (range of 52-2052)
Population: Safety Analysis Set
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Enzalutamide
Number analyzed (Participants) | 67
Days | 168 [58 to 581]

25. Secondary Outcome: Time to PSA Progression
Description: Time to PSA progression is defined as the time interval from the first study drug dose to the first date of PSA progression. PSA progression is defined as a ≥ 25% increase in PSA with an absolute increase of ≥ 2 ng/mL above the nadir unless the PSA next measurement(s), if available, does not confirm the PSA progression.
Time Frame: From first dose until the EOS date of 27-Apr-2017; median duration of treatment of 1666.0 days (range of 52-2052)
Population: Safety Analysis Set
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Enzalutamide
Number analyzed (Participants) | 67
Days | NA [NA to NA] — Could not be estimated due to the low number of events

26. Secondary Outcome: PSA Doubling Time
Description: PSA doubling time was to be calculated from the slope estimated from a linear regression of the natural log of PSA fitted on time, if the slope was positive. Since the slope was negative for all participants, PSA doubling time could not be calculated.
Time Frame: From Baseline to Week 25
Population: Safety Analysis Set with a positive PSA versus time slope
Arm/Group | Enzalutamide
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30 days after last dose of study drug; median duration of treatment of 1666.0 days (range of 52-2052)
Arm/Group | Enzalutamide
All-Cause Mortality (participants affected / at risk) | 5/67
Serious Adverse Events (participants affected / at risk) | 24/67
Other Adverse Events (participants affected / at risk) | 66/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzalutamide (N=67)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 2 (2)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 4 (4)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1)
Chronic fatigue syndrome (General disorders) | 1 (1)
Device dislocation (General disorders) | 1 (1)
General physical health deterioration (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Metastases to abdominal cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Normal pressure hydrocephalus (Nervous system disorders) | 1 (1)
Seizure anoxic (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Prostatic calcification (Reproductive system and breast disorders) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzalutamide (N=67)
Abdominal discomfort (Gastrointestinal disorders) | 4 (5)
Constipation (Gastrointestinal disorders) | 9 (11)
Diarrhoea (Gastrointestinal disorders) | 11 (14)
Dry mouth (Gastrointestinal disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 11 (14)
Fatigue (General disorders) | 28 (40)
Oedema peripheral (General disorders) | 8 (10)
Cystitis (Infections and infestations) | 4 (4)
Nasopharyngitis (Infections and infestations) | 6 (9)
Pneumonia (Infections and infestations) | 5 (6)
Fall (Injury, poisoning and procedural complications) | 4 (5)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (12)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 7 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (9)
Dizziness (Nervous system disorders) | 5 (5)
Headache (Nervous system disorders) | 4 (8)
Memory impairment (Nervous system disorders) | 6 (7)
Depression (Psychiatric disorders) | 5 (5)
Breast pain (Reproductive system and breast disorders) | 6 (7)
Gynaecomastia (Reproductive system and breast disorders) | 36 (43)
Nipple pain (Reproductive system and breast disorders) | 13 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Hot flush (Vascular disorders) | 15 (18)
Hypertension (Vascular disorders) | 17 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data.Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.